CLINICAL TRIAL: NCT07336550
Title: AFFAP Trial: The Comparative Evaluation of Audit and Feedback-based De-implementation Strategies to Reduce Low-value Prescribing in Primary Care in Patients Over 65 Years of Age.
Brief Title: Reduction of Low-value Prescribing Through Audit and Feedback
Acronym: AFFAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Collaborators: Biobizkaia (Unknown); Health Department of the Basque Government (Unknown); European Union (Other); Carlos III Health Institute (ISCIII), Spain (Unknown)
Responsible Party: Principal Investigator, Mikel Baza Bueno, Principal Investigator, Basque Health Service
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024111054; 2018111085 (Other Grant/Funding Number: Health Department of the Basque Government); 2021111024 (Other Grant/Funding Number: Health Department of the Basque Government); PI21/00025 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII) and European Union (European Regional Development Fund "A way to make Europe")); RD24/0005/0017 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII) and European Union); RD21/0016/0003 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII) and European Union (NextGenerationEU funds, MRR)); RD16/0007/0002 (Other Grant/Funding Number: Instituto de Salud Carlos III (ISCIII) and European Union (European Regional Development Fund "A way to make Europe"))
Record Dates: First submitted 2025-12-17; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Inappropriate Prescribing; Implementation Science; Behavioral Sciences
Keywords: low-value pharmacological prescription; De-implementation; Stepped-wedge design; Benzodiazepines; Proton pump inhibitors; Opioids; audit and feedback

STUDY DESIGN:
Intervention Model Description: A closed-cohort stepped-wedge cluster-randomised trial will be conducted. All health centre clusters will start under the control condition, and at each step, three centres will be randomly assigned to crossover to the intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): All health centre clusters will start under the control condition
  Interventions: Behavioral: Usual AF
- Intervention (Experimental): At each step, three centres will be randomly assigned to crossover to the intervention
  Interventions: Behavioral: Usual AF; Behavioral: Facilitated AF

INTERVENTIONS:
Behavioral: Usual AF — The strategy currently used as a management tool to evaluate healthcare performance focusing on processes and outcomes, as part of Osakidetza's operating contract: provision of AF, sent to PC centres every 4 months with data on overall rates of PIP, lists of patients over 65 years old who have a potentially inappropriate prescription of at least one of the drugs of interest, and provision of support materials related to appropriate prescribing and recommendations on deprescribing.
Behavioral: Facilitated AF — Based on a facilitation component delivered by PC pharmacy staff. Specifically, the PC pharmacists will conduct a facilitation session with the centre's clinicians in which they will review the magnitude of PIP in the centre (PIP rates), appropriateness/inappropriateness criteria, and guidelines to encourage deprescribing, and draw up an action plan at clinician and centre levels.
  Arms: Intervention

SUMMARY:
The objective is to estimate the effect attributable to a primary care pharmacist-led audit and feedback (AF) strategy compared to the currently used AF strategy as a management tool to evaluate healthcare performance focusing on processes and outcomes, for reducing the rate of patients over 65 years of age with potentially inappropriate prescribing (PIP) of benzodiazepines, proton pump inhibitors and opioids.

A closed-cohort stepped-wedge cluster-randomised trial will be conducted in nine PC centres from Barakaldo-Sestao Integrated Health Organization, Basque Health Service (Osakidetza). All health centre clusters will start under the control condition, and at each step, some three centres will be randomly assigned to crossover to the intervention, under which they will be exposed to an additional component of AF, namely, primary care pharmacist-led facilitation.

Mixed-methods analysis will be performed, gathering quantitative data to assess the results of the implementations at health centre and clinician levels, and qualitative data to assess the feasibility and perceived impact of the de-implementation strategies from the clinicians' perspective, and explore the experience and satisfaction of patients regarding the healthcare received.

This study will provide useful knowledge on the effect attributable to a more intensive AF strategy (facilitated AF) compared to standard procedures of AF reports, and of the characteristics of AF that are most effective.

ELIGIBILITY:
PRIMARY CARE CENTERS IN THE BARAKALDO-SESTAO INTEGRATED HEALTHCARE ORGANISATION OF OSAKIDETZA-BASQUE HEALTH SERVICE:

Inclusion Criteria:

* collaboration is achieved from at least 51% of the General Practitioners (GP) or at least 4 GPs
* At least 60 patients aged 65 years or older on at least one of the drugs of interest that may be potentially inappropriately prescribed

Exclusion Criteria:

* N/A

PATIENTS ASSIGNED TO THE PARTICIPATING PC CENTERS:

Inclusion Criteria:

* Patients over 65 years of age with any of the following unsuitability criteria:
* PIP of benzodiazepines: patients on benzodiazepines for more than 3 months
* PIP of proton pump inhibitors: patients on proton pump inhibitors for more than 8 weeks without a diagnosed gastrointestinal disease and with no long-term prescription of gastrotoxic drugs.
* PIP of opioids: patients on opioids for non-cancer pain for more than 3 months.

Exclusion Criteria:

* Patients who, in the opinion of the general practitioner, are not suitable candidates for tapering or discontinuation of the potentially inappropriately prescribed drug
* Patients residing in care homes
* Patients receiving palliative care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Primary effectiveness: Proportion of patients with deprescribing or tapering of any of the PIP | From baseline to 16 months
  proportion of patients for whom appropriateness is achieved, either through deprescribing or tapering (for example, dose reduction) of any of the drugs potentially inappropriately prescribed in the patients included in the clusters.

SECONDARY OUTCOMES:
Secondary effectiveness: Proportion of patients with deprescribing or tapering for each PIP | From baseline to 16 months
  proportion of patients in whom appropriateness is achieved for each of the potentially inappropriately prescribed drugs assessed separately
Secondary Effectiveness: Rate of new PIP | From baseline to 16 months
  Rate of new PIP among patients over 65 years old seeking medical care during the study period
Adoption: Percentage of General Practitioners who agree to receive the active components of the strategies | From baseline to 16 months
  Percentage of doctors, out of the total number invited to participate at the start of the intervention, who agree to receive the active components of the strategies, as well as the characteristics of those who do and do not agree to participate.
Degree of implementation fidelity | From baseline to 16 months
  The degree of fidelity with which each strategy has been implemented compared to what was originally planned will be evaluated. For this, the implementation process and any adaptations made to the strategies or their active components will be recorded and subsequently described. Furthermore, we will evaluate the degree of exposure of GPs to the strategies.
General Practitioners´ perception of the feasibility and acceptability | From baseline to 22 months
  GPs perception of the feasibility and acceptability of the deprescribing strategy based on the AF to adapt/reduce their practice of unnecessary pharmacological prescribing.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Research Unit of Bizkaia, Barakaldo, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that support future results will be shared, after deidentification
Supporting Information: Study Protocol
Time Frame: Starting 6 months after the publication of results
Access Criteria: Since data supporting the present study will mostly concern routine data retrieved from the electronic health record of the Basque Health Service-Osakidetza, it will only be made available on reasonable request to the study guarantors (proposals should be directed to the Responsible Party). It will only be shared with researchers whose proposed use of the data has been approved by an independent review committee identified for this purpose.